CLINICAL TRIAL: NCT07041411
Title: Histological and Radiological Evaluation of Crosslinked vs Not Cross Linked Graft in Transcretal Sinus Elevation in Severely Resorbed Maxilla. A Prospective, Controlled Study
Brief Title: Transcrestal Sinus Lift With OSSIX Bone vs BIOSS Collagen
Acronym: TSL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo (Other)
Responsible Party: Principal Investigator, Luigi Canullo, prof, Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dontiart
Record Dates: First submitted 2025-05-22; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Sinus Lift; Graft Materials; Transcrestal Approach

STUDY DESIGN:
Intervention Model Description: controlled clinical investigation
Who Masked: Outcomes Assessor
Masking Description: assessors analyzed blindly receiving anonymized bone samples and CBCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSSIX Bone (Experimental): OSSIX® Bone in the maxillary sinus elevation.
  Interventions: Procedure: maxillary sinus elevation through transcrestal approach using OSSIX® Bone
- Bio-Oss collagen (Active Comparator): Bio-Oss Collagen in the maxillary sinus elevation.
  Interventions: Procedure: maxillary sinus elevation through transcrestal approach using OSSIX® Bone

INTERVENTIONS:
Procedure: maxillary sinus elevation through transcrestal approach using OSSIX® Bone — After a careful radiologic analysis, using a surgical guide, maxillary sinus elevation through transcrestal access to sinus mucosa was achieved. The elevation of the maxillary sinus mucosa was performed through micro-elevators and graft material was inserted.
  Other Names: maxillary sinus elevation through transcrestal approach using Bio-Oss® Bone; Ossix Bone

SUMMARY:
Primary: Histologically analyse the quality of bone regeneration after graft material insertion in severely resorbed maxilla.

Secondary: Radiological analysis of the volume of the bone regenerations with the shirnkage rate of the graft material. clinical study of 20 patients 13 in OSSIX Bone group 13 in Bio-Oss Collagen group all patients requiring a regenerative procedure (sinus lift) having less than 3mm of residual bone height (RBH) with the impossibility to place the implants at the time of regenerative proc 6 months follow up for the first endpoint. (collection of the histological sample) 12 months follow up - long term clinical evaluation. tests performed: Cone Beam Computed Tomography (CBCT), clinical evaluation, X-ray

DETAILED DESCRIPTION:
Visit 1 - Screening Visit - preoperative visit (informed consent, dental mouth cleaning, CBCT, intraoral scanning).

Visit 2 - Baseline visit - T0 (surgical procedure) Sinus elevation with OSSIX® Bone or Bio-Oss® Collagen, periapical x-ray, intraoral photo with microscope.

Visit 3 - Follow up visit - 14 days - suture removal, clinical evaluation and patient satisfaction questionnaire.

Visit 4 - Follow up visit - 180days (One week before) Cone Beam Computed Tomography (CBCT), Dental mouth cleaning, intraoral scanning.

(Second surgery) implant site preparation and histological sample collection, implant placement, insertion torque value, implant stability, peri-apical x-ray, intraoral scanning and photography.

Visit 5 - Follow up visit - 194 days suture removal and clinical evaluation. Visit 6 - Follow up visit - 270 days Implant stability, clinical examination, definitive restoration and periapical x-ray Visit 7- Follow up visit - 365 days Implant stability, peri-apical x-ray, definitive restoration, Cone Beam Computed Tomography (CBCT), intraoral scanning and picture.

ELIGIBILITY:
Inclusion criteria:

1. Patient requiring vertical elevation of the maxillary sinus.
2. Residual alveolar bone height of edentulous maxilla below the floor of the maxillary sinus of < 3-4 mm.
3. Males and females between 30-80 years old
4. Patients with healthy periodontal conditions (Treated periodontitis, Plaque Index (PI) <25%, Bleeding on Probing (BoP) <25%).
5. Patients that are willing to sign an informed consent and participate in a clinical Study.
6. Generally fit and healthy and able to undergo oral surgical procedures under local anesthesia.
7. Teeth at the surgical site which required removal were extracted a minimum of 12 weeks prior to sinus floor elevation.

Exclusion criteria:

1. Patient requiring vertical elevation of the maxillary sinus with native bone crest height > 5 mm
2. Patients who smoke over 5 cigarettes/day
3. Pregnancy (confirmed by verbal inquiry)
4. Chronic systemic pathologies (e.g. diabetes) and neoplastic of the Oro-Facial District 4.
5. Patients taking bisphosphonates
6. Any sites where an implant already failed sites
7. Untreated Periodontitis
8. Dental sites with acute infections
9. Chronic inflammatory diseases of the oral cavity
10. Autoimmune diseases (cortisone intake)
11. Allergy declared to one or more medicaments to be used during treatment
12. Alcoholics patients and/or drug addicts
13. Patients with known collagen hypersensitivity.
14. Patients with sensitivity to porcine-derived materials.
15. History or malignant tumors of the maxillary sinus
16. History of local radiation therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2025-03-22 (Actual)

PRIMARY OUTCOMES:
histological analysis | 6 months after graft insertion
  samples were collected and histologically and immunohistologically analyzed

SECONDARY OUTCOMES:
radiological analyis | 12 months
  preoperatively Cone Beam Computed Tomography (CBCT) was compared to 12 months CBCT. The volume of bone regeneration was measured by performing a semi-automatic segmentation using a specific segmentation software (3D Slicer) and measured in mm3.

CONTACTS AND LOCATIONS:
Locations (1):
- Studi Odontoiatrici Luigi Canullo, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No
data will be shared if required